CLINICAL TRIAL: NCT02702752
Title: Dynamic Changes in Stromal Cell-derived Factor-1α Levels in Acute and Stabilized Heart Disease - ACUTE MYOCARDIAL INFARCTION, ATRIAL FIBRILLATION, AND HEART FAILURE (THE DYNASDY STUDY)
Brief Title: Dynamic Changes in SDF-1α Levels in Acute and Stabilized Heart Disease
Acronym: DYNASDY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Lawkesh Vimal Hurry, M.D., Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-15007626
Record Dates: First submitted 2015-11-15; First posted 2016-03-09 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Atrial Fibrillation; Ischemic Heart Disease; Congestive Heart Failure
Keywords: Heart diseases stromal differentiation factor alpha 1
MeSH Terms: conditions — Atrial Fibrillation; Myocardial Ischemia; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DYNASDY (Other): The study considers changes in SDF-1α levels in response to treatment of cardiac disease (myocardial infarction, heart failure or atrial fibrillation). SDF-1α levels will be measured at the acute stages of the disease, after stabilization and at longer term as detailed below. Levels of SDF-1α will be correlated to the outcome of disease.
  Interventions: Other: DYNASDY
- Control group (Active Comparator): A control group of 20 subjects without cardiac disease (including hypertension), diabetes, hypercholesterolemia, and malignant disease.
  Interventions: Other: DYNASDY

INTERVENTIONS:
Other: DYNASDY — Measurement of SDF-1 alpha levels i patients' blood samples.

SUMMARY:
The aims of the present study are to measure dynamic changes over time in the plasma level of SDF-1α in patients with confirmed diagnoses of AMI, AF and CHF and in so doing:

1. Monitor the plasma level of SDF-1α at the diagnosis, during and after the long term treatment of AMI, AF and CHF. The SDF-1α level of patients is expected to decrease during treatment of the aforementioned conditions.
2. Correlate the plasma level of SDF-1α in relation to clinical, biochemical characteristics of Acute Myocardial Infarction(AMI), Atrial Fibrillation(AF) and Congestive Heart Failure (CHF). In so doing, the investigators expect that SDF-1α will correlate with the severity of heart disease.
3. Study the dynamic of SDF-1α pertaining to its property as prognostic indicator for the long term follow up risk of readmission and mortality of patients diagnosed with AMI, AF or CHF.

DETAILED DESCRIPTION:
The study considers changes in SDF-1α levels in response to treatment of cardiac disease (myocardial infarction, heart failure or atrial fibrillation). SDF-1α levels will be measured at the acute stages of the disease, after stabilization and at longer term as detailed below. Levels of SDF-1α will be correlated to the outcome of disease.

BLOOD SAMPLING AND MEASUREMENT OF SDF-1Α A blood sample of about 5 ml will be sampled by peripheral venepuncture and anticoagulated with heparin. Blood samples will be spun for 15 minutes at 1000g within 30 minutes of collection. The resulting plasma will be stored at -80°C until analysis. Levels of SDF-1α in the plasma will be determined using a commercially available ELISA kit according to the manufacturer's instructions.

Analyses will be performed at the Clinical Research Centre, Copenhagen University Hospital Hvidovre.

PATIENTS Patients are included from the in-patient department of the Department of Cardiology, Hvidovre University Hospital. Patients are eligible for inclusion if diagnosed with myocardial infarction, atrial fibrillation or heart failure, provided they do not suffer from malignant disease, diabetes mellitus types I or II and have a life expectancy of at least one year.

Exclusion criteria are based upon the fact that serum SDF-1α levels are elevated in malignant diseases as SDF-1α contributes to neoangiogenesis of the tumour mass, and SDF-1α levels have recently been demonstrated to be elevated in diabetes.

The investigators will include 20 patients with each of the cardiac conditions mentioned as well as a control group of 20 subjects without cardiac disease (including hypertension), diabetes, hypercholesterolemia, and malignant disease.

PATIENTS WITH MYOCARDIAL INFARCTION Patients presenting with non-ST elevation myocardial infarction (NSTEMI) are included. The diagnostic criteria are symptoms of cardiac ischaemia (angina or angina-equivalent symptoms) and elevated troponin T (above 14 ng/mL) and/ or ECG changes of ischemia (horizontal or downsloping ST depression ≥ 0.5 mm at the J-point in ≥ 2 contiguous leads).

Patients are excluded if they are diagnosed with a "type 2 myocardial infarction", i.e. myocardial ischaemia due to mismatch between myocardial oxygen demand and supply due to conditions such as severe anaemia, arrhythmia or hypotension. Patients are also excluded if they are not referred for coronary angiography, if they have atrial fibrillation or if they have cardiac failure with LVEF ≤ 40%.

The SDF-1α levels of patients will be measured on the first day of hospitalization, after coronary angiography, before discharge (approximately day 3-5), and three months after inclusion.

PATIENTS WITH ATRIAL FIBRILLATION Patients presenting with ECG-documented atrial fibrillation are included if unstable, i.e. if heart rate exceeds 100 and in-patient treatment is indicated. Patients are excluded if they suffer from unstable ischaemic heart disease (unstable angina or myocardial infarction), heart failure with LVEF ≤ 40% or if the arrhythmia is secondary to another condition such as an infection.

SDF-1α levels will be measured on the first day of the hospitalization, at the time of discharge (after medical or electrical cardioversion or after stabilization of the heart rate) and three months after inclusion.

PATIENTS WITH CONGESTIVE HEART FAILURE Patients are included if presenting with decompensated heart failure. They must have symptoms of heart failure (dyspnoea and/ or oedema) severe enough to warrant in-patient treatment. The diagnosis must be confirmed by echocardiography showing LVEF ≤ 40%. Patients are excluded if suffering from unstable ischaemic heart disease (unstable angina or myocardial infarction) or atrial fibrillation.

The SDF-1α levels of will be measured on the first day of the hospitalization, after medical stabilization at the time of discharge, and three months after inclusion.

PATIENT INCLUSION AND DATA COLLECTION Patient inclusion will take place during three consecutive months. Patients are included within the first day of hospital admittance. Each day, members of the project group will screen all patients admitted within the last day and personally contact those eligible for inclusion. Patients will be informed verbally and given the written participant information. Patients will be given time for consideration and if they accept participation, they will be asked to sign the consent form. Due to the project design, according to which the first blood samples are to be taken within the first day of hospitalization, patients are asked to consent to project participation on the day of initial contact with the research group member. Conversations will be held in a private setting in the department, and patients are invited to bring relations, if they so prefer.

As regards the control group, these will be included from patients initially referred for outpatient evaluation at the Department of Cardiology, but in whom no cardiac disease is found. Members of the project group will screen the patients in the Outpatients Department and personally contact those eligible for inclusion in the control group. The control group will be selected so as to be age-matched with the patients. Information about the project will be provided as for the patients.

Based upon information in the patients' medical files, it will be registered whether patients suffer from hypertension, peripheral vascular disease, stroke, transient cerebral ischaemia, chronic obstructive pulmonary disease or renal insufficiency.

Medication at time of admittance to hospital and medication given during the hospitalization will be registered. Clinical status (dyspnoea, palpitations, oedema, blood pressure and heart rate) at the time of inclusion and at the time discharge from hospital will be noted. This information will be sought from patient files and the Kiso system used for recording vital parameters in patients.

The recorded information (pre-existing conditions, medication and clinical status at the two time-points) will be available for the project group. This information will be used for background demographics, in the evaluation of how levels of SDF-1α correlate to clinical status, and to allow for correction of factors, such as medication, on the levels of SDF-1α.

FOLLOW-UP All patients are expected to be seen in the Outpatients' Department 2-3 months after discharge from hospital. This appointment is part of the standard treatment and control plan for patients with AF, CHF and NSTEMI, respectively and not arranged as a part of the project. Certain information will be registered from the patient files at the time of follow-up: Clinical status (NYHA class, oedema, pulmonary congestion, and angina), heart rhythm, medication, and any intercurrent hospital admissions.

One year after inclusion, patient files will be reviewed and the following information registered: Whether the patient is alive and any cardiovascular rehospitalisation. In the case of hospitalization, the date of admission, duration and diagnosis will be registered. Statistical considerations and data analysis Baseline data of SDF-1α levels and patient demographics (including comorbidities and use of medication) will be evaluated using descriptive statistics. Normally distributed data will be presented as mean and standard deviation, whereas skewed data will be presented as median and range. If necessary, skewed data will be transformed.

The influence of patient characteristics (such as age, sex and comorbidities) on SDF-1α levels will be evaluated using multiple regression analysis with SDF-1α level as dependent variable and patient characteristics as explanatory variables. SDF-1α levels will be compared between the patient groups using analysis of variance (ANOVA).

Within each group of patients, the changes in SDF-1α levels over time (three time points) will be analysed using ANOVA.

The investigators have previously measured SDF-1α levels in patients with various types of AF (permanent versus paroxysmal). Based upon these results (SDF-1α levels and standard deviations in the different groups), the investigators have estimated that the proposed sample size of 20 patients in each disease group will confer the study sufficient statistical power.

The statistical analyses will be performed in collaboration with statistician Steen Ladelund (Clinical Research Centre, Hvidovre University Hospital).

THE RESEARCH GROUP

The study will be conducted in close collaboration between the Department of Cardiology and the Clinical Research Centre at Hvidovre University Hospital. The research group will consist of the following persons:

Dr L. Vimal Hurry, MD, is project responsible. He is a junior doctor at the Department of Cardiology and doing research work beside his clinical employment.

Dr Ulrik Dixen, MD, PhD, is a consultant at the Department of Cardiology. Dr Ulrik Dixen has conducted AF research for several years and is experienced in planning and conducting clinical studies, as well as in supervising junior researchers.

Dr Nadia Landex, MD, PhD, is training in cardiology, currently at Roskilde University Hospital. She did her PhD in histochemistry and has used her experience in basic research to initiate research in biomarkers in AF at Hvidovre University Hospital, including research topic, project planning and the initial laboratory work.

Medical student Maha Alsawaf has written her bachelor thesis in the cardiology research group and has basic research experience. Maha Alsawaf will assist with inclusion of the patients.

Medical student Ema Rastoder is experienced in clinical research and skilled in patient communication. Ema Rastoder will assist with inclusion of patients.

Project members from the Clincial Research Centre are:

Head of Department Ove Andersen, MD, PhD, who has extensive experience in biomarker research at all stages from project development to implementation of research results.

Anne Langkilde, MSc, PhD, is likewise experienced in biomarker research, particularly in the prognostic importance of biomarkers in disease. Anne Langkilde has been a close collaborator in the initial projects regarding measurement of biomarkers in AF.

Together, the research team has experience of biomarker research as well as access to research laboratory with highly skilled laboratory technicians.

ELIGIBILITY:
Inclusion Criteria:

Patients are included from the in-patient department of the Department of Cardiology, Hvidovre University Hospital. Patients are eligible for inclusion if diagnosed with one of the following diseases:

* myocardial infarction
* atrial fibrillation
* heart failure

Exclusion Criteria: Patients must not suffer from one of the follwing conditions:

* malignant disease
* diabetes mellitus types I or II
* have a life expectancy of at least one year.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-12 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Dynamic changes in SDF-1α levels for use as a prognostic factor during and after treatment of Acute Myocardial Infarction, Atrial Fibrillation and Heart Failure. | 6 months
  This study aims to evaluate the dynamic changes in SDF-1α levels during and after treatment of three major heart diseases. Results will aid in the understanding of the role of SDF-1α in cardiac disease. If disease progression and treatment effect is reflected in the levels of SDF-1α, measurement of this biomarker will be a valuable tool for monitoring disease course and treatment effect and, in so doing, help in risk evaluation and individualized treatment of patients suffering from cardiac disease.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Landex, Ph.D., Study Chair — Department of Cardiology, Roskilde University Hospital; Ema Ema Rastoder, MB, Study Chair — Department of Cardiology, Copenhagen University Hospital Hvidovre; Maha Maha Alsawaf, MB, Study Chair — Department of Cardiology, Copenhagen University Hospital Hvidovre; Anne Langkilde, MS, Ph.D., Study Director — Clinical Research Centre, Copenhagen University Hospital Hvidovre; Ove Andersen, M.D., Ph.D., Study Director — Clinical Research Centre, Copenhagen University Hospital Hvidovre
Locations (1):
- Copenhagen University Hospital Hvidovre, Hvidovre, Capital Region of Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No
It a randomized study where all data will be anonymous.